CLINICAL TRIAL: NCT01724567
Title: Copenhagen Study of Obese Patients With Ischemic Heart Disease Undergoing Low Energy Diet or Interval Training: A Randomized Clinical Trial
Brief Title: Copenhagen Study of Obese Patients With Ischemic Heart Disease Undergoing Low Energy Diet or Interval Training
Acronym: CUT-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eva Prescott (Other)
Collaborators: University of Copenhagen (Other); Amager Hospital (Other); Bispebjerg Hospital (Other); Copenhagen University Hospital at Herlev (Other); Copenhagen University Hospital, Hvidovre (Other); Rigshospitalet, Denmark (Other); University of California, Davis (Other); Texas A&M University (Other); University of Aarhus (Other)
Responsible Party: Sponsor-Investigator, Eva Prescott, MD, MDsc, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CUT-IT
Record Dates: First submitted 2012-10-26; First posted 2012-11-12 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Ischemic Heart Disease; Obesity
Keywords: Interval Training; Weight Loss; Secondary Prevention; Rehabilitation; Cardiovascular Risk Factors
MeSH Terms: conditions — Myocardial Ischemia; Obesity; Weight Loss | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weight Loss (Experimental): 12 weeks of Low Calorie Diet to obtain a 10 - 15 % weight loss. Followed by 40 weeks on a weight maintenance diet and interval training 2 times a week.
  Interventions: Other: Weight Loss
- Interval Training (Experimental): 12 weeks of interval training 3 times a week followed by 40 weeks of interval training 2 times a week.
  Interventions: Other: Interval Training

INTERVENTIONS:
Other: Interval Training — Interval training (IT) on an exercise bike 3 times a week, for the first 12 weeks, followed by 40 weeks of IT 2 times a week on exercise bike. Each training session consists of active intervals with a total duration of 16 minutes (durations intervals between 1 and 4 minutes) at 90% of maximal heart rate. Active intervals are separated by active pauses at 60% of maximal heart rate.
  Arms: Interval Training
Other: Weight Loss — Low calorie diet approx. 1000 kcal/day for 8 - 10 weeks to obtain a 10 - 15 % weight loss.
  Arms: Weight Loss

SUMMARY:
The purpose of the study is to make a head-to-head comparison of weight loss and interval training as methods of secondary prevention in overweight patients with ischemic heart disease.

DETAILED DESCRIPTION:
In western countries 80 % of patients with ischemic heart disease (IHD) are overweight (BMI > 25). Weight loss using a low energy diet (LED, 800 - 1000 kcal/day) has been shown to induce a considerable weight loss in obese but otherwise healthy patients and to reduce the risk of cardiovascular disease and diabetes in these subjects. Additionally, a British study using a very low energy diet (VLED, 600 kcal/day) to obtain weight loss, has shown that subject with diagnosed type 2 diabetes had their blood glucose normalized after an 8 week VLED. However, the effect of LED has never been examined in overweight patients with IHD.

Several studies have shown that patients with IHD have a beneficial effect of exercise training regarding mortality and reduction in cardiovascular risk factors. A Norwegian group has shown that aerobic interval training results in the biggest increase in maximal oxygen uptake (VO2max). A high VO2max is correlated to decreased mortality in patients with IHD.

In conclusion, weight loss and exercise are known strategies in preventing progression of IHD and development of type 2 diabetes in these patients, however a head-to-head comparison of the two methods has never been made and it is unknown which intervention is the most effective in improving cardiovascular risk profile. Furthermore, several mechanisms behind the known beneficial effect of these interventions are unknown.

ELIGIBILITY:
Inclusion Criteria:

* Stable Ischemic Heart Disease
* BMI 28 - 40 kg/m2

Exclusion criteria:

* Known Diabetes Mellitus
* Repeated Fasting plasma glucose ≥ 7 mmol/L or Hba1c > 7 %
* Severe or moderate valve disease
* Main stem stenosis
* Severe heart failure, Ejection Fraction < 35 %
* Physical or mental disability which are expected to prevent completion of intervention
* Severe Chronic obstructive Pulmonary Disease (COPD) (FEV1 < 50 % of expected) or asthma
* Active cancer
* Severe kidney (GFR < 40 ml/hour) or severe liver disease
* Severe ischemia or arrhythmias during exercise test
* 2. or 3. degree atrio-ventricular (AV) block, not protected by pacemaker
* Organised training more than 2 times a week prior to inclusion
* Significant weight loss or weight gain (> 5 %)3 month prior to inclusion
* Not able to comprehend written and oral informed consent
* Hormone treatment

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in Coronary Flow Reserve following the diet or training intervention and a maintenance period | 0, 12 and 52 weeks
  Assessed by a non-invasive echocardiographic Doppler measurement

SECONDARY OUTCOMES:
Change in Heart Rate Variability and silent ischemia following the diet or training intervention and a maintenance period | 0, 12 and 52 weeks
  Assessed by Holter Monitoring for 24 - 48 hours
Change in endothelial function following the diet or training intervention and a maintenance period | 0, 12 and 52 weeks
  Using the Endopat 2000 from Itamar
Change in systolic and diastolic function following the diet or training intervention and a maintenance period | 0, 12 and 52 weeks
  Assessed by echocardiography resting and during physiological and medical stress.
Change in body composition following the diet or training intervention and a maintenance period | 0, 12 and 52 weeks
  Assessed by anthropometry, dual X-ray absorptiometry (DXA) (lean body mass, percentage adipose tissue) and abdominal MRI (liver fat, muscle fat, subcutaneous fat and visceral fat at the level of L3).
Change in myocardial blood flow following the diet or training intervention and a maintenance period | 0, 12 and 52 weeks
  Assessed by positron emission tomography of the heart
Change in insulin action, beta cell function and incretin secretion following the diet or training intervention and a maintenance period | 0, 12 and 52 weeks
  A Oral Glucose Tolerance Test is performed.
Change in oxidized lipids and lipoprotein particle size following the diet or training intervention and a maintenance period | 0, 12 and 52 weeks
Change in peak oxygen uptake (VO2max) following the diet or training intervention and a maintenance period | 0, 12 and 52 weeks
  Assessed using a bicycle ergometer
Change in blood pressure following the diet or training intervention and a maintenance period | 0, 12 and 52 weeks
Change in inflammatory markers in urin, blood and adipose tissue following the diet or training intervention and a maintenance period | 0, 12 and 52 weeks
Change in quality of life following the diet or training intervention and a maintenance period | 0, 12 and 52 weeks
Change in ceramides, diacylglycerol og endocannabinoid (CB)-1 receptors in adipose tissue following the diet or training intervention and a maintenance period | 0, 12 and 52 weeks
Change in hormones derived from adipose tissue following the diet or training intervention and a maintenance period | 0, 12 and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eva Prescott, MD, DMsc, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

REFERENCES:
- [Background] Pedersen LR, Olsen RH, Frederiksen M, Astrup A, Chabanova E, Hasbak P, Holst JJ, Kjaer A, Newman JW, Walzem R, Wisloff U, Sajadieh A, Haugaard SB, Prescott E. Copenhagen study of overweight patients with coronary artery disease undergoing low energy diet or interval training: the randomized CUT-IT trial protocol. BMC Cardiovasc Disord. 2013 Nov 19;13:106. doi: 10.1186/1471-2261-13-106. PMID 24252596
- [Background] Pedersen LR, Olsen RH, Jurs A, Astrup A, Chabanova E, Simonsen L, Wisloff U, Haugaard SB, Prescott E. A randomised trial comparing weight loss with aerobic exercise in overweight individuals with coronary artery disease: The CUT-IT trial. Eur J Prev Cardiol. 2015 Aug;22(8):1009-17. doi: 10.1177/2047487314545280. Epub 2014 Jul 31. PMID 25082954
- [Derived] Pedersen LR, Olsen RH, Anholm C, Astrup A, Eugen-Olsen J, Fenger M, Simonsen L, Walzem RL, Haugaard SB, Prescott E. Effects of 1 year of exercise training versus combined exercise training and weight loss on body composition, low-grade inflammation and lipids in overweight patients with coronary artery disease: a randomized trial. Cardiovasc Diabetol. 2019 Oct 1;18(1):127. doi: 10.1186/s12933-019-0934-x. PMID 31575375
- [Derived] Pedersen LR, Olsen RH, Anholm C, Walzem RL, Fenger M, Eugen-Olsen J, Haugaard SB, Prescott E. Weight loss is superior to exercise in improving the atherogenic lipid profile in a sedentary, overweight population with stable coronary artery disease: A randomized trial. Atherosclerosis. 2016 Mar;246:221-8. doi: 10.1016/j.atherosclerosis.2016.01.001. Epub 2016 Jan 13. PMID 26803431
- [Derived] Pedersen LR, Olsen RH, Jurs A, Anholm C, Fenger M, Haugaard SB, Prescott E. A randomized trial comparing the effect of weight loss and exercise training on insulin sensitivity and glucose metabolism in coronary artery disease. Metabolism. 2015 Oct;64(10):1298-307. doi: 10.1016/j.metabol.2015.07.007. Epub 2015 Jul 17. PMID 26296452
- [Derived] Olsen RH, Pedersen LR, Jurs A, Snoer M, Haugaard SB, Prescott E. A randomised trial comparing the effect of exercise training and weight loss on microvascular function in coronary artery disease. Int J Cardiol. 2015 Apr 15;185:229-35. doi: 10.1016/j.ijcard.2015.03.118. Epub 2015 Mar 11. PMID 25802037